CLINICAL TRIAL: NCT05577858
Title: Effect of a Pulse-based USDA-diet on Gut Microbial Metabolites and Biomarkers of Healthspan: A 18-week Randomized Controlled Crossover Feeding Study in Older Adults
Brief Title: Protein-Distinct Macronutrient-Equivalent Diet 1
Acronym: PRODMED1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Responsible Party: Principal Investigator, Moul Dey, Professor, South Dakota State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2209011-EXP
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Healthy Lifestyle

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Blinding will be implemented to the extent possible. A researcher, unaware of the study goals and not involved with downstream data analyses will use a 1:1 block randomization to allocate participants to the diets in the first arm. Food service personnel (care provider) will not be aware of study goals and allocations. Metabolomic assays will be run in a blinded manner.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meat based (Other): Animal protein-based dietary intervention
  Interventions: Other: Meat based
- Pulse based (Experimental): Pulse-protein-based dietary intervention
  Interventions: Other: Pulse based

INTERVENTIONS:
Other: Meat based — Omnivorous diet following dietary guidelines
  Arms: Meat based
Other: Pulse based — Lacto-ovo-vegetarian pulse-based diet following dietary guidelines
  Arms: Pulse based

SUMMARY:
Plant-based diets are naturally low in Methionine (Met), and also low in precursor molecules (e.g L-carnitine, choline, betaine, etc.) producing microbiota-mediated proatherogenic TMAO. Among plant proteins, pulses are rich in micronutrients, and dietary fibers, making them ideal for microbiome-stimulating, nutrient-dense, healthful dietary patterns. However, daily pulse intake remains low at 8% in America despite recommendations by DGA, a resource to guide health promotion across communities. A significant body of preclinical data, waiting to be translated to humans, suggests that dietary Met restriction can trigger beneficial metabolic and anti-inflammatory adaptations leading to improved chronic health and longevity. The central hypothesis is that a pulse-protein-based healthy diet can be simultaneously equivalent to omnivorous diets in protein content and yet naturally lower in Met and TMAO to improve glycemic control, body composition, and immunometabolic flexibility to reduce the risk of chronic diseases and improve healthspan. The goal is to systematically elucidate for the first time the effects of a lacto-vegetarian feeding pattern with pulses as the primary protein source on a comprehensive panel of ~500 traditional and next-generation biomarkers of health, and assess the role of the gut microbiota in mediating such effects. We also aim to interrogate the potential concern about the lower bioavailability of non-heme iron from pulses.

ELIGIBILITY:
Inclusion Criteria:

* Generally good health status based on routine physical in the past 12 months, current healthy status
* Normal HbA1C, not underweight
* Age 60 years or more, all races, both sexes and all education level
* Do not have any special dietary requirements and willing to consume vegetarian diet
* Willingness to comply with the study protocol, including on-site meal consumption and sample/data collection.

Exclusion Criteria:

* Probiotic, long-term antibiotic, and tobacco/drug/alcohol use
* Not on any special diet within 3 months of recruitment
* Impaired kidney functions
* Active history of cancer, diabetes, heart, liver, and kidney diseases
* Major gastrointestinal disorders in the past 3 months
* History of heart attacks or stroke
* Unable to meet in-person visit requirements for dining, picking up meals, and tests
* Any mental health condition that would affect the ability to provide written informed consent.
* If they had not had a routine health checkup during the 12 months prior to recruitment.
* If they were unwilling to abstain from taking certain nutritional supplements, alcohol, or non-study foods during the study period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Ferritin | 16 weeks
  Microplate assay
Concentration of TMAO in blood | 16 weeks
  Using LC/MS based method method
Fasting blood glucose concentration in blood | 16 weeks
  Using Glucometer

SECONDARY OUTCOMES:
Body weight in kilograms | 16 weeks
  Measurement
Concentration of CRP in blood | 16 weeks
  Microplate assay
Gut microbiota composition and diversity | 16 weeks
  16S rRNA gene sequencing
Fat and lean mass in kg using DXA for body composition measures | 16 weeks
  DEXA scan
Concentration of sulfur containing amino acids in blood | 16 weeks
  LC/MS based method
Digestible indispensable amino acid score using different amino acid concentrations | 16 weeks
  Using standard equation
Concentration of IGF-1 in blood | 16 weeks
  Using Microplate assay kit
Concentration of IGF-BP3 in blood | 16 weeks
  Using Microplate assay kit
Concentration of Fasting insulin in blood | 16 weeks
  Using Microplate assay kit
Peak heights of several complex lipids panel using metabolomics technique | 16 weeks
  LC/MS based assay
Concentration Short-chain fatty acid panel in stool | 16 weeks
  using LC/MS based assay
Peak heights of several Biogenic amines panel using metabolomics technique | 16 weeks
  using LC/MS based assay
Muscle strength using Isokinetic muscle testing | 16 weeks
  Biodex ergometer
Balance assessment using balance | 16 weeks
  Mechanography
Grip force per kg mass | 16 weeks
  using Dynamometer
Blood pressure in mm Hg | 16 weeks
  Upper arm cuff

CONTACTS AND LOCATIONS:
Overall Officials: Moul Dey, Ph.D., Principal Investigator — South Dakota State University
Locations (1):
- South Dakota State University, Wagner Hall 416, Brookings, South Dakota, United States

REFERENCES:
- [Derived] de Vargas BO, Vaezi S, Freeling JL, Zhang Y, Weidauer L, Lee CL, Zhao J, Dey M. Design and Implementation of the Protein-Distinct Macronutrient-Equivalent Diet (PRODMED) Study: An Eighteen-Week Randomized Crossover Feeding Trial Among Free-Living Rural Older Adults. Curr Dev Nutr. 2025 Mar 24;9(5):104588. doi: 10.1016/j.cdnut.2025.104588. eCollection 2025 May. PMID 40291832